CLINICAL TRIAL: NCT01370382
Title: Comparison Between the New Highly Sensitive Troponin T and the Conventional Troponin T Test of the 4th Generation for the Early Identification of Myocardial Necrosis in Elderly Patients With Acute Coronary Syndromes Without ST-segment Elevation
Brief Title: Comparison Between the New Highly Sensitive Troponin T and the Conventional Troponin T Test in Elderly Patients
Acronym: BOSCH2
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Klinikum Nürnberg (Other)
Responsible Party: Principal Investigator, Philipp Bahrmann, MD, University of Erlangen-Nürnberg Medical School
Other Study IDs: BOSCH2
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Acute Coronary Syndrome
Keywords: geriatrics; troponin; electrocardiography; diagnosis; myocardial infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Disease; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Time interval: Patients are divided according to the interval between the onset of chest pain symptoms and presentation at the hospital in an "early"(<4 hours) and "late"(> = 4 hours) group.

SUMMARY:
The planned cohort study shall clarify whether the use of biomarkers leads to improved diagnostic assessment of elderly patients. The study will evaluate the clinical value of biomarkers (highly sensitive Troponin T, Troponin T of the 4th generation) in elderly patients. These biomarkers are analyzed together with the symptoms and other parameters collected at admission. The diagnosis of myocardial infarction could be made earlier and more accurately with the help of biomarkers, in particular the highly sensitive troponin T.

DETAILED DESCRIPTION:
All consecutive patients with acute symptoms and an age over 70 years will be recruited for the study during 6 months. Medical history, physical examination, vital signs including heart rate, blood pressure, body temperature, and any concomitant diseases are raised on admission in the Emergency Department. Blood samples are taken for determination of routine laboratory. Highly sensitive troponin T is determined as part of the routine. Troponin T is measured from the same blood sample with a conventional test of the 4th generation. A second blood sample is taken as part of routine 4-6 hours after the onset of symptoms to confirm or rule out any acute coronary syndrome. Patients are divided according to the interval between the onset of symptoms and presentation at the hospital in an "early"(<4 hours) and "late"(> = 4 hours) group.

The Barthel Index as a geriatric assessment is raised. An electrocardiogram is written in all patients at recording and evaluated. An echocardiographic examination is performed in all patients for measurement of heart valve function, left ventricular diameter, ejection fraction (LVEF) and diastolic function to differentiate into other mechanisms for the release of troponin. According to the results of the echocardiographic examination, patients are divided into sub-groups (LV-EF> = 55%) and without preserved ejection fraction (LVEF <55%). The recording physician estimates after receiving the results of the investigations and routine laboratory whether a myocardial infarction or heart failure is present. He subsequently makes the decision about further treatment. The medical records will be evaluated after completion of the stay in hospital by two experienced cardiologists, whether a heart attack, heart failure or other disease was present. High sensitivity Troponin T and Troponin T of the 4th generation are compared for the early and correct diagnosis of acute coronary syndrome.

Objectives:

1. Incidence of acute coronary syndromes without ST-segment elevation in elderly patients by using the highly sensitive biomarker troponin T,
2. Comparison with the incidence of acute coronary syndromes without ST-segment elevation in the same group by the use of troponin T of the 4th generation
3. Survey on differential diagnoses such as heart failure or other cardiac diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 or older
* Signed informed consent

Exclusion Criteria:

* Hospitalization for unstable angina pectoris within the last 2 month
* ST-segment elevation myocardial infarction
* Heart valve defects with need for surgical intervention
* Coronary bypass surgery or percutaneous transluminal angioplasty within the last 3 months
* Planned elective coronary revascularization
* Serum creatinine> 2.0 mg / dl (177 µmol / liter)
* Serum potassium> 5.5 mmol / l Limited survival probability within the next 3 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Emergency department of the Klinikum Nürnberg (50,000 attendances per year; the department caters to an urban population of approximately 1 million).
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of acute coronary syndromes without ST-segment elevation during hospitalization. | 30 days

SECONDARY OUTCOMES:
Accurate diagnosis of myocardial infarction (without knowledge of biomarkers) | 30 days
Accurate diagnosis of acute heart failure (without knowledge of biomarkers) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Bahrmann, MD, Principal Investigator — Department of Internal Medicine II-2, Institute for Biomedicine of Ageing, Friedrich-Alexander-University Erlangen-Nürnberg
Locations (1):
- Klinikum, Nuremberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bahrmann P, Heppner HJ, Christ M, Bertsch T, Sieber C. Early detection of non-ST-elevation myocardial infarction in geriatric patients by a new high-sensitive cardiac troponin T assay. Aging Clin Exp Res. 2012 Jun;24(3):290-4. doi: 10.3275/7927. Epub 2011 Sep 26. PMID 21952408
- [Result] Bahrmann P, Christ M, Bahrmann A, Rittger H, Heppner HJ, Achenbach S, Bertsch T, Sieber CC. A 3-hour diagnostic algorithm for non-ST-elevation myocardial infarction using high-sensitivity cardiac troponin T in unselected older patients presenting to the emergency department. J Am Med Dir Assoc. 2013 Jun;14(6):409-16. doi: 10.1016/j.jamda.2012.12.005. Epub 2013 Jan 30. PMID 23375478
- [Result] Bahrmann P, Bahrmann A, Breithardt OA, Daniel WG, Christ M, Sieber CC, Bertsch T. Additional diagnostic and prognostic value of copeptin ultra-sensitive for diagnosis of non-ST-elevation myocardial infarction in older patients presenting to the emergency department. Clin Chem Lab Med. 2013 Jun;51(6):1307-19. doi: 10.1515/cclm-2012-0401. PMID 23314553